CLINICAL TRIAL: NCT06273774
Title: A Multiple Dose Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MK-8189 in Participants With Bipolar I Disorder
Brief Title: A Study of MK-8189 in Participants With Bipolar I Disorder (MK-8189-020)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 8189-020; MK-8189-020 (Other: MSD)
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — MK-8189

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Panel A: 24 mg MK-8189 (Experimental): Participants received 24 mg MK-8189 once daily (QD) for 14 days.
  Interventions: Drug: MK-8189
- Panel B: 16 & 24 mg MK-8189 (Experimental): Participants received 16 mg MK-8189 QD on Days 1 to 3 and 24 mg MK-8189 QD on Days 4 to 14.
  Interventions: Drug: MK-8189
- Panel C: 8, 16, & 24 mg MK-8189 (Experimental): Participants received 8 mg MK-8189 Day 1, 16 mg on Day 2 ,and 24 mg on QD Days 3 to 14.
  Interventions: Drug: MK-8189
- Panel C: Placebo (Placebo Comparator): Participants received Panel C MK-8189-matching placebo QD for 14 days.
  Interventions: Drug: Placebo
- Panel A: Placebo (Placebo Comparator): Participants received Panel A MK-8189-matching placebo QD for 14 days.
  Interventions: Drug: Placebo
- Panel B: Placebo (Placebo Comparator): Participants received Panel B MK-8189-matching placebo for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8189 — Oral Tablet
  Arms: Panel A: 24 mg MK-8189; Panel B: 16 & 24 mg MK-8189; Panel C: 8, 16, & 24 mg MK-8189
Drug: Placebo — Oral Tablet
  Arms: Panel A: Placebo; Panel B: Placebo; Panel C: Placebo

SUMMARY:
The goal of this study is to evaluate the safety and tolerability of MK-8189 in participants with stable bipolar I disorder. There was no hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Meets diagnostic criteria for bipolar I disorder, manic or mixed features according to the Diagnostic and statistical manual of Mental Disorders TR (DSM-5 TR) and considered to be in a non-acute phase of their illness.
* History of receiving and tolerating antipsychotic medication within the usual dose range employed for bipolar I disorder.
* Body mass index is 18 and 40 kg/m^2, inclusive.
* If currently taking an antipsychotic, is able to discontinue use at least 5 days prior to study start and the duration of the study.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Untreated or uncompensated endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases.
* Evidence or history of a primary DSM-5 axis I psychiatric diagnosis other than those specified for inclusion.
* History of cancer (malignancy).
* Evidence or history of mental retardation, borderline personality disorder, or organic brain syndrome.
* History of neuroleptic malignant syndrome or moderate to severe tardive dyskinesia.
* Substance-induced psychotic disorder or behavioral disturbance.
* DSM-5 TR defined substance use disorder within 3 months of screening.
* History of seizure disorder beyond childhood or is receiving treatment with any anticonvulsant to prevent seizures.
* Positive test(s) for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus.
* Major surgery or donation/loss of 1 unit of blood within 4 weeks prior to screening.
* Received any vaccine starting from 30 days prior to study intervention or is scheduled to receive any vaccine through 30 days following study intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Woodland International Research Group-Clinical Research ( Site 0009), Little Rock, Arkansas
  - Atlanta Center for Medical Research ( Site 0001), Atlanta, Georgia
  - Hassman Research Institute Marlton Site ( Site 0006), Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After the safety and tolerability was reviewed from the first cohort of Panel A, a protocol amendment was written to give the option to enroll either Panel B or Panel C. Panel C was selected to be enrolled; no participants were enrolled in Panel B and no data was collected for this panel.
Groups:
- Panel B: 16 & 24 mg MK-8189: Participants received 16 mg MK-8189 QD on Days 1 to 3 and 24 mg MK-8189 QD on Days 4 to 14. No participants were enrolled in Panel B.
- Panel B: Placebo: Participants received Panel B MK-8189 matching placebo on days 1-14. No participants were enrolled in Panel B.
- Panel C: 8, 16, & 24 mg MK-8189: Participants received 8 mg MK-8189 Day 1, 16 mg on Day 2, and 24 mg on QD Days 3 to 14.
- Panel C Placebo: Participants received Panel C MK-8189-matching placebo QD for 14 days.
Period: Overall Study
Arm/Group | Panel A: 24 mg MK-8189 | Panel A: Placebo | Panel B: 16 & 24 mg MK-8189 | Panel B: Placebo | Panel C: 8, 16, & 24 mg MK-8189 | Panel C Placebo
Started (No participants were enrolled in Panel B.) | 12 | 5 | 0 | 0 | 13 | 4
Completed | 12 | 5 | 0 | 0 | 12 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Participant was out of state. | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Panel B and no data was collected for this panel.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: 24 mg MK-8189 | Panel A: Placebo | Panel C: 8, 16, & 24 mg MK-8189 | Panel C Placebo | Total
Number analyzed (Participants) | 12 | 5 | 13 | 4 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (11.5) | 40.8 (11.9) | 43.1 (12.6) | 51.5 (10.0) | 43.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 3 | 16
  Male | 8 | 2 | 7 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 0 | 5
  Not Hispanic or Latino | 10 | 3 | 11 | 4 | 28
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 10 | 1 | 18
  White | 7 | 3 | 2 | 3 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 28 days
Population: All participants who received at least one dose of treatment were included in the analysis. No participants were enrolled in Panel B and no data was collected for Panel B. One participant in Panel C receiving 24 mg MK-8189 experienced an adverse event and was down-titrated to 12 mg MK-8189 per protocol.
Measure: Number; unit: Participants
Groups:
- Panel A: MK-8189 24 mg: Participants received 24 mg of MK-8189 once daily (QD) for 14 days.
- Panel C: MK-8189 8 mg: Participants received 8 mg of MK-8189 on Day 1.
- Panel C: 16 mg MK-8189: Participants received 16 mg of MK-8189 on Day 2.
- Panel C: MK-8189 24 mg: Participants received 24 mg of MK-8189 on Days 3 to 14. One participant received 24 mg of MK-8189 on Days 3-8 and then was titrated down to 12 mg for Days 9-14 due to an AE.
- Panel C: MK-8189 12 mg: Participant was down-titrated per protocol to 12 mg of MK-8189 for Days 9 through 14.
- Panel C: Placebo: Participants received MK-8189-matching placebo QD for up to 14 days.
Arm/Group | Panel A: MK-8189 24 mg | Panel A: Placebo | Panel B: 16 & 24 mg MK-8189 | Panel B: Placebo | Panel C: MK-8189 8 mg | Panel C: 16 mg MK-8189 | Panel C: MK-8189 24 mg | Panel C: MK-8189 12 mg | Panel C: Placebo
Number analyzed (Participants) | 12 | 5 | 0 | 0 | 13 | 13 | 13 | 1 | 4
Participants | 9 | 4 |  |  | 1 | 4 | 6 | 0 | 1

2. Primary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: as for outcome 1
Time Frame: Up to 14 days
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Panel C: MK-8189 16 mg: Participants received 16 mg of MK-8189 on Day 2.
Arm/Group | Panel A: MK-8189 24 mg | Panel A: Placebo | Panel B: 16 & 24 mg MK-8189 | Panel B: Placebo | Panel C: MK-8189 8 mg | Panel C: MK-8189 16 mg | Panel C: MK-8189 24 mg | Panel C: MK-8189 12 mg | Panel C: Placebo
Number analyzed (Participants) | 12 | 5 | 0 | 0 | 13 | 13 | 13 | 1 | 4
Participants | 3 | 1 |  |  | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days.
Description: All-Cause Mortality is reported for all randomized participants. Serious Adverse Events and Other Adverse Events are reported for all participants who received treatment. No participants were enrolled in Panel B and no data was collected for Panel B. One participant in Panel C receiving 24 mg MK-8189 experienced an adverse event and was down-titrated to 12 mg MK-8189 per protocol. AEs were reported separately for this participant at the 12 mg dose.
Arm/Group | Panel A: MK-8189 24 mg | Panel A: Placebo | Panel C: MK-8189 8 mg | Panel C: MK-8189 16 mg | Panel C: MK-8189 24 mg | Panel C: MK-8189 12 mg | Panel C: Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5 | 0/13 | 0/13 | 0/13 | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/5 | 0/13 | 0/13 | 0/13 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 9/12 | 4/5 | 1/13 | 4/13 | 6/13 | 0/1 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-8189 24 mg (N=12) | Panel A: Placebo (N=5) | Panel C: MK-8189 8 mg (N=13) | Panel C: MK-8189 16 mg (N=13) | Panel C: MK-8189 24 mg (N=13) | Panel C: MK-8189 12 mg (N=1) | Panel C: Placebo (N=4)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-8189 24 mg (N=12) | Panel A: Placebo (N=5) | Panel C: MK-8189 8 mg (N=13) | Panel C: MK-8189 16 mg (N=13) | Panel C: MK-8189 24 mg (N=13) | Panel C: MK-8189 12 mg (N=1) | Panel C: Placebo (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oromandibular dystonia (Nervous system disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT06273774/Prot_SAP_000.pdf